CLINICAL TRIAL: NCT01787968
Title: Congenital Transmission of Lineages I and II of Trypanosoma Cruzi
Status: Completed | Type: Observational
Sponsor: Tulane University School of Public Health and Tropical Medicine (Other)
Collaborators: Institute for Clinical Effectiveness and Health Policy (Other); Université Libre de Bruxelles (Other); Instituto de Enfermedades Infecciosas y Parasitol Antonio Vidal (Unknown); Lab de Parasitologia Universidad Autonoma de Yucatan (Unknown)
Responsible Party: Principal Investigator, Dr. Pierre Buekens, W.H. Watkins Professor and Dean, Tulane University School of Public Health and Tropical Medicine
Organization: Tulane University (Other)
Other Study IDs: R01AI083563 (NIH)
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Chagas Disease
Keywords: Congenital transmission; Trypanosoma cruzi; Chagas disease
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, blood with guanidine, dry spots on filter papers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TcI, TcII: TcI: T. cruzi seropositive mothers from countries where TcI predominates, or/and with TcI genotyping TcII: T. cruzi seropositive mothers from countries where TcII (non-TcI) predominates, or/and with TcII (non-TcI) genotyping

SUMMARY:
T. cruzi has been divided into two main lineages: T. cruzi I (TcI) and T. cruzi II (TcII, including all non-TcI). TcI is predominant in Mexico and Central America, while TcII (non-TcI) is predominant in most of South America, including Argentina. In recent studies from Argentina, the risk of congenital transmission has been estimated to vary between 2.6 percent and 7.9 percent. By contrast, we know very little about the congenital transmission of TcI. It has been suggested that congenital transmission of T. cruzi is strain related, and there is an urgent need to know if TcI transmits differently than TcII (non-TcI). Our primary hypothesis is that congenital transmission rates are different for TcI versus TcII. Our secondary hypothesis is that the characteristics of T. cruzi infected mothers (e.g., age, parity, transmission in previous pregnancies) and their exposure to vectors are different in regions where TcI is predominant versus regions where TcII (non-TcI) is predominant. To test these hypotheses, we propose to conduct a prospective study to enroll at delivery 13,000 women in Mexico, 7,500 women in Honduras, and 10,000 women in Argentina. We will measure transmitted maternal T. cruzi antibodies in cord blood, and, if the results are positive, we will identify infants who are congenitally infected by performing parasitological examinations on cord blood and at 4-8 weeks, and serological follow-up at 10 months. We will also perform standard PCR, real-time quantitative PCR, and T. cruzi genotyping on maternal blood, standard PCR and T. cruzi genotyping on the cord blood of congenitally infected newborns, and serological examinations on siblings. We will estimate the exposure to vectors in the household. In addition, we will measure prenatal outcomes among infected and uninfected infants with seropositive mothers, and the birth weight of their siblings. The specific aims of this study are: 1) To determine the rate of congenital transmission of TcI compared to TcII (non-TcI); 2) To compare the T. cruzi infected mothers' characteristics and exposure to vectors in regions where TcI is predominant and regions where TcII (non-TcI) is predominant; and 3) To describe the birth outcomes of infected and uninfected infants born to TcI and TcII seropositive women.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old or more, informed consent, live birth.

Exclusion Criteria:

* Women residing outside of the follow-up area.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women delivering in participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 28348 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Congenital transmission of Trypanosoma cruzi | Two years
  We will identify infants who are congenitally infected by performing parasitological examinations on cord blood, on venous blood at 4-8 weeks, and serological follow-up at 10 months. Standard PCR, quantitative real-time PCR (qPCR), and T. cruzi genotyping will be performed on maternal blood and cord blood.

SECONDARY OUTCOMES:
Birth outcomes | Two years
  Perinatal outcomes (premature rupture of the membranes, birthweight, gestational age, IUGR, and neonatal complications) will be measured among infected and uninfected infants with seropositive mothers, and birthweight will be measured among infected and uninfected siblings.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Buekens, MD, PhD, Principal Investigator — Tulane SPHTM
Locations (5):
- Tulane School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States
- Institute for Clinical Effectiveness and Health Policy, Buenos Aires, Argentina
- Laboratory of Parasitology, Universite Libre de Bruxelles, Brussels, Belgium
- Inst. de Enfermedades Infecciosas y Parasitol Antonio Vidal, Tegucigalpa, Honduras
- Lab. de Parasitologia, Universidad Autonoma de Yucatan, Mérida, Mexico

REFERENCES:
- [Derived] Buekens P, Cafferata ML, Alger J, Althabe F, Belizan JM, Carlier Y, Ciganda A, Dumonteil E, Gamboa-Leon R, Howard E, Matute ML, Sosa-Estani S, Truyens C, Wesson D, Zuniga C. Congenital transmission of Trypanosoma cruzi in Argentina, Honduras, and Mexico: study protocol. Reprod Health. 2013 Oct 11;10:55. doi: 10.1186/1742-4755-10-55. PMID 24119247
- See also: Related Info — http://www.chagascongenito.info/